CLINICAL TRIAL: NCT04864782
Title: A Study of QL1604 Plus Chemotherapy in Subjects With Stage IVB, Recurrent, or Metastatic Cervical Cancer
Brief Title: QL1604 Plus Chemotherapy in Subjects With Stage IVB, Recurrent, or Metastatic Cervical Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Phase 2 completed, phase 3 sponsor decided to terminate
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1604-301
Record Dates: First submitted 2020-12-04; First posted 2021-04-29 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — spartalizumab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1604+Chemotherapy (Experimental): On Day 1 of each 21-day cycle, participants receive an intravenous (IV) infusion of QL1604 200 mg plus Investigator choice of chemotherapy (paclitaxel 175 mg/m^2 plus cisplatin 70 mg/m^2 or paclitaxel 175 mg/m^2 plus carboplatin Area Under the Curve (AUC) 6)
  Interventions: Drug: QL1604; Drug: Paclitaxel injection; Drug: Cisplatin/Carboplatin

INTERVENTIONS:
Drug: QL1604 — Intravenous Infusion
  Other Names: PD-1 monoclonal antibody
Drug: Paclitaxel injection — Intravenous Infusion
Drug: Cisplatin/Carboplatin — Intravenous Infusion

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PD-1 Inhibitor (QL1604) plus chemotherapy in patients with Stage IV, recurrent, or metastatic cervical cancer. Possible chemotherapy regimens include: paclitaxel plus cisplatin and paclitaxel plus carboplatin.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts.The first stage is a single-arm clinical trial, and the second stage is a controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years
2. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Life expectancy of at least 12 weeks.
4. At least one measurable lesion (according to RECIST v1.1)
5. Cervical squamous cell carcinoma, adenocarcinoma and adenosquamous cell carcinoma diagnosed by histopathology and confirmed by imaging as recurrent or stage ⅣB cervical cancer.
6. No brain metastasis, or no meningeal metastasis.
7. Patients must have normal function as defined:

   1. ANC≥1.5*10^9/L; PLT≥90*10^9/L, Hb≥90 g/L,
   2. Total Bilirubin (TBIL)≤1.5*Upper Limit of Normal(ULN), Alanine Transaminase (ALT)and Aspartate Aminotransferase(AST)≤2.5*ULN.For liver metastasis patients, ALT and AST≤5*ULN,
   3. Cr≤ 1.5*ULN, or creatinine clearance rate ≥50 mL/min,
   4. Proteinuria <2+，if proteinuria≥ 2+ and 24 hours total urine protein < 1.0 g
   5. LVEF≥ 50%.
8. Any unresolved AEs ≤ CTCAE Grade 1 (except alopecia).
9. Negative pregnancy test for females of child-bearing potentials.
10. Patients with reproductive function agreed to take effective contraceptive measures during the treatment and in 6 months after the end of administration.
11. Patients must be able to understand and volunteer to sign the informed consent.

Exclusion Criteria:

1. Has received more than 2 courses of palliative chemotherapy for treatment of cervical cancer.
2. Has received prior chemoradiotherapy within 3 months before enrollment,or has received prior radiotherapy within 2 weaks before enrollment.
3. Has received prior surgery therapy within 2 weaks before enrollment,or has not recovered from the effects of surgery therapy.
4. Is currently participating in or has participated in a study of an investigational agent within 4 weeks before enrollment.
5. Has any active autoimmune diseases or a history of autoimmune diseases (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid hyperfunction; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adulthood; asthma patients who require bronchodilators for medical intervention cannot be included).
6. Is using immunosuppressive agents or systemic hormonal therapy to achieve immunosuppressive purposes (agents amount > 10 mg / day of prednisone or other therapeutic hormones), and continue to use within 2 weeks before enrollment.
7. Known history of hypersensitivity to macromolecular protein preparation or any components of the QL1604 formulation, or any components of the study drugs.
8. Has uncontrolled clinically significant cardiac and cerebral vascular diseases within 6 months before enrollment, including but not limited to the following: myocardial infarction, severe or unstable angina, coronary artery/peripheral artery bypass grafting, congestive heart failure, cerebrovascular accident (including transient ischemic attack).
9. Symptomatic congestive heart failure (New York Heart Association Grade II-IV), or NCI-CTCAE v5.0 ≥ 2 arrhythmia, atrial fibrillation of any grade, or clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention.
10. Has active infection or an unexplained fever > 38.5°C during screening visits( subjects with tumor fever may be enrolled at the discretion of the investigator).
11. Hepatitis b surface antigen (HBsAg) positive and/or hepatitis b core antibody (HBcAb) positive and HBVDNA>103copies/ml, hepatitis c virus antibody positive .
12. Known history of human immunodeficiency virus (HIV) infection, or other acquired or congenital immunodeficiency diseases,or has a history of organ transplantation (except corneal transplantation).
13. Has been vaccinated with live anti-tumor vaccine, or have received anti-tumor immunotherapy, or may receive other systemic anti-tumor treatments during the study period.
14. Peripheral neuropathy≥ CTCAE Grade 2.
15. History of psychotropic substance abuse, alcoholism or drug abuse.
16. Has a clear history of neurological or mental disorders, including epilepsy or dementia.
17. Patients with other malignancies witnin 5 years( except cured basal cell carcinoma of skin cancer, papillary thyroid carcinoma).
18. At the discretion of the investigator, there are patients with serious concomitant disease that compromises patient safety or affects the patient's completion of the study,such as unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 160 mmHg, diastolic blood pressure > 110 mmHg), serious diabetes, thyroid diseases, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with adverse events | Up to 90 days from last dose
  The incidence and severity of adverse events (AE),serious adverse events (SAE) and treatment-emergent adverse events (TEAEs) according to CTCAE V5.0
Objective response rate (ORR) as assessed by investigator based on RECIST v1.1 and iRECIST | approximately 2 years
  Objective response rate (ORR) as assessed by investigator based on RECIST v1.1 and iRECIST

SECONDARY OUTCOMES:
Progression-free survival (PFS) as assessed by investigator based on RECIST v1.1 and iRECIST | approximately 2 years
  Progression-free survival (PFS) is defined as time from the date of randomization to the date of first documentation of disease progression or death due to any cause(whichever occurs earlier)
Overall survival(OS) | approximately 2 years
  Overall survival(OS) is defined as the time from randomization to death due to any cause
Duration of response(DOR) | approximately 2 years
  Duration of response(DOR) as assessed by investigator based on RECIST v1.1 and iRECIST
Time to progress (TTP) | approximately 2 years
  Time to progress (TTP) as assessed by investigator based on RECIST v1.1 and iRECIST
AUC of QL1604 | approximately 1 years
  Area under curve from zero to infinity
Cmax of QL1604 | approximately 1 years
  Peak concentration
Cmin of QL1604 | approximately 1 years
  The trough value at steady state
Tmax of QL1604 | approximately 1 years
  Time to Cmax
T1/2 of QL1604 | approximately 1 years
  Half life
Vss of QL1604 | approximately 1 years
  Steady-state apparent volume of distribution based on plasma concentration
CLT(total body clearance) of QL1604 | approximately 1 years
  Total body clearance
Immunogenicity | approximately 1 years
  The titer of anti-drug antibodies (ADA)and neutralizing antibodies(Nab)

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangzhou, China